CLINICAL TRIAL: NCT05725005
Title: A Phase 1, Open-label, Positron Emission Tomography Study in Healthy Subjects to Determine the Relationship Between Plasma Concentration and Target Occupancy of ASN51 Following Repeated Oral Doses
Brief Title: PET Study of Repeated ASN51 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Asceneuron S.A. (Industry)
Collaborators: Hammersmith Medicines Research (Other); Invicro (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: ASN51-103
Record Dates: First submitted 2022-12-30; First posted 2023-02-13 (Actual); Results first posted 2025-05-08 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: ASN51 Low Dose (Experimental): Participants received low dose of ASN51, orally, once-daily (QD) for 14 days in fasted or fed state.
  Interventions: Drug: ASN51
- Group 2: ASN51 High Dose (Experimental): Participants received high dose of ASN51, orally, QD for 14 days in fasted or fed state.
  Interventions: Drug: ASN51

INTERVENTIONS:
Drug: ASN51 — Oral capsule

SUMMARY:
This is a phase 1, open-label, dose escalation, positron emission tomography (PET) study to investigate the brain occupancy of O-GlcNAcase, and the pharmacodynamics (PD) response in peripheral blood mononuclear cells (PBMCs), after repeated doses of ASN51 in healthy participants.

DETAILED DESCRIPTION:
The clinical data from the first-in-human single- and multiple-ascending dose study of ASN51 (ASN51-101), and the adaptive-design PET study of O-GlcNAcase brain ASN51 occupancy after single oral doses (ASN51-102), showed acceptable safety, tolerability and pharmacokinetics (PK). However, to date, no assessment of receptor occupancy (RO) after multiple doses of ASN51 and at plasma concentrations below the EC50 have been done. Hence, the purpose of this study is to assess brain O-GlcNAcase RO using PET following repeated doses of ASN51. The study will also characterise the PBMC response (including the effect of food), and further assess the safety, tolerability, PK, and PK/RO relationship, after repeated ASN51 doses.

The results of this study will be used to select doses for subsequent studies in participants.

ELIGIBILITY:
Inclusion Criteria:

1. Normotensive male volunteer (PET participants).
2. Male or female volunteer of non-childbearing potential (PBMC-only participants).
3. Deemed healthy on the basis of a clinical history, physical and neurological examination, electrocardiogram (ECG), vital signs, and laboratory tests of blood and urine.
4. Agree to follow the contraception requirements of the trial.
5. Able to give fully informed written consent.

Exclusion Criteria:

1. Significant (> 10%) recent weight change.
2. Positive tests for hepatitis B and hepatitis C, human immunodeficiency virus (HIV).
3. Severe adverse reaction to any drug.
4. Sensitivity to trial medication.
5. Drug or alcohol abuse.
6. Regular consumption of xanthine-containing products.
7. Frequent use of nicotine-containing products.
8. Severe adverse reaction to any drug.
9. Sensitivity to trial medication (all participants) or PET imaging radioligand (PET participants).
10. Use of over-the-counter medication (with the exception of paracetamol [acetaminophen]) during the 7 days before the first dose of radioligand (PET participants) or trial medication (PBMC participants) (or longer if the medicine is a potential enzyme inducer), or prescribed medication during the 28 days before first dose of radioligand (PET participants) or trial medication (PBMC participants).
11. Received vaccine against severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) within 2 weeks of screening.
12. Participation in other clinical trials of unlicensed medicines.
13. Loss of more than 400 milliliters (mL) blood, within the 3 months before the first dose of tracer (PET participants) or trial medication (PBMC participants).
14. Clinically relevant abnormal findings at the screening assessment, including ECG abnormalities (all participants) or those identified by MRI scan (PET participants only).
15. Acute or chronic illness.
16. Clinically relevant abnormal history of or concurrent medical (including neurological or psychiatric) condition.
17. Positive columbia-suicide severity rating scale (C-SSRS) result.
18. Vegan.
19. Possibility that volunteer will not cooperate.
20. Unsatisfactory venous access.
21. Objection by general practitioner (GP).
22. PET participants only: significant exposure to research related radiation (more than 10 millisievert [mSv]) within the previous 12 months.
23. Contraindications to arterial cannulation (e.g., allen's test indicates risk) or magnetic resonance imaging (MRI) scanning (e.g., presence of a cardiac pacemaker or other implanted electronic device or a history of claustrophobia).

Ages: 22 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2023-01-26 (Actual); Primary Completion 2023-04-04 (Actual); Study Completion 2023-06-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adeep Puri, MD, Principal Investigator — Hammersmith Medicines Research
Locations (1):
- Hammersmith, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at an investigative site in the United Kingdom from 26 January 2023 to 08 June 2023.
Groups:
- Group 1: ASN51 Low Dose: Participants received low dose of ASN51, orally, once daily (QD), for 14 days in fasted or fed state.
Period: Overall Study
Arm/Group | Group 1: ASN51 Low Dose | Group 2: ASN51 High Dose
Started | 6 | 6
PET Population (Positron emission tomography (PET) population included all participants in the safety population who had a baseline PET scan, at least 1 post-baseline PET scan, and a pharmacokinetic (PK) result immediately preceding a PET scan.) | 4 | 4
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received at least one dose of the study drug.
Groups:
- Group 1: ASN51 Low Dose: Participants received low dose of ASN51, orally, QD for 14 days in fasted or fed state.
- Total: Total of all reporting groups
Arm/Group | Group 1: ASN51 Low Dose | Group 2: ASN51 High Dose | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.2 (7.68) | 37.3 (6.12) | 38.8 (6.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 6 | 6 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 6 | 12
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 3 | 4
  White | 5 | 2 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Protein O-GlcNAcylation in Peripheral Blood Mononuclear Cells (PBMCs)
Description: Protein O-GlcNAcylation in PBMCs at different time-point is reported.
Time Frame: Pre-dose on Days 1, 2, 11, and 14; 8 hours post-dose on Day 1, 11 and 14; 12 hours post-dose on Day 1 and 14, 24 hours post-dose on Day 15; 72 hours post-dose on Day 17; 144 hours post-dose on Day 20
Population: Pharmacodynamics (PD) analysis population included all participants in the safety population for who a PBMC measure is available. Number analyzed is the number of participants evaluated in respective arm at a specified timepoint.
Measure: Mean (Standard Deviation); unit: percentage of protein O-GlcNAcylation
Arm/Group | Group 1: ASN51 Low Dose | Group 2: ASN51 High Dose
Number analyzed (Participants) | 6 | 6
percentage of protein O-GlcNAcylation
  Pre-dose on Day 1 | 100.0 (0.00) | 100.0 (0.00)
  8 hours post-dose on Day 1 | 219.33 (74.728) | 232.79 (94.193)
  12 hours post-dose on Day 1 | 291.02 (117.673) | 190.48 (56.442)
  Pre-dose on Day 2 | 183.83 (84.144) | 188.02 (96.636)
  Pre-dose on Day 11: number analyzed (Participants) | 2 | 2
  Pre-dose on Day 11 | 205.70 (19.045) | 188.30 (126.761)
  8 hours post-dose on Day 11 | 302.19 (49.840) | 346.01 (233.011)
  Pre-dose on day 14 | 196.42 (99.330) | 197.54 (98.510)
  8 hours post-dose on Day 14 | 297.01 (119.672) | 282.51 (151.609)
  12 hours post-dose on Day 14 | 303.24 (147.572) | 305.26 (167.261)
  24 hours post-dose on Day 15 | 166.19 (62.638) | 160.38 (58.879)
  72 hours post-dose on Day 17 | 169.66 (45.654) | 192.67 (128.801)
  144 hours post-dose on Day 20 | 168.68 (40.767) | 187.14 (126.539)

2. Primary Outcome: Regional Total Volume of Distribution (VT) of [18F]-IMA601 in Frontal Lobe at Each Brain Scan
Description: Regional VT of [18F]-IMA601 in frontal lobe at each brain scan was measured with a PET scan. Participants received an intravenous (IV) dose of the radiolabelled tracer, [18F]-IMA601, at the start of each PET scan. Participant wise data was reported for this outcome measure.
Time Frame: PET Scan 1 (Baseline), PET Scan 2 (post-dose on Day 1), PET Scan 3 (Day 4 [for participants 1, 2 (Group 2 only) 3, and 4 (Group 1 only)] and Day 9 [for participant 2 in Group 1 only] and Day 10 [for participant 4 in Group 2 only]) after final ASN51 dose
Population: PET population included all participants in the safety population who had a baseline PET scan, at least 1 post-baseline PET scan, and a PK result immediately preceding a PET scan. Here, "number analyzed" signifies specific participant evaluated in respective arm at a specified timepoint.
Measure: Number; unit: milliliters/cubic centimeter(mL/cm^3)
Arm/Group | Group 1: ASN51 Low Dose | Group 2: ASN51 High Dose
Number analyzed (Participants) | 4 | 4
milliliters/cubic centimeter(mL/cm^3)
  Participant 1, PET Scan 1, Baseline: number analyzed (Participants) | 1 | 1
  Participant 1, PET Scan 1, Baseline | 11.47 | 15.91
  Participant 1, PET Scan 2, Day 1: number analyzed (Participants) | 1 | 1
  Participant 1, PET Scan 2, Day 1 | 1.97 | 1.60
  Participant 1, PET Scan 3, Day 4: number analyzed (Participants) | 1 | 1
  Participant 1, PET Scan 3, Day 4 | 2.68 | 3.67
  Participant 2, PET Scan 1, Baseline: number analyzed (Participants) | 1 | 1
  Participant 2, PET Scan 1, Baseline | 14.81 | 13.53
  Participant 2, PET Scan 2, Day 1: number analyzed (Participants) | 1 | 1
  Participant 2, PET Scan 2, Day 1 | 2.02 | 2.46
  Participant 2, PET Scan 3, Day 4: number analyzed (Participants) | 0 | 1
  Participant 2, PET Scan 3, Day 4 |  | 2.91
  Participant 2, PET Scan 3, Day 9: number analyzed (Participants) | 1 | 0
  Participant 2, PET Scan 3, Day 9 | 16.81 |
  Participant 3, PET Scan 1, Baseline: number analyzed (Participants) | 1 | 1
  Participant 3, PET Scan 1, Baseline | NA — Data was not reported as the PET scan findings failed to converge a meaningful VT. | 17.34
  Participant 3, PET Scan 2, Day 1: number analyzed (Participants) | 1 | 1
  Participant 3, PET Scan 2, Day 1 | 2.20 | 1.56
  Participant 3, PET Scan 3, Day 4: number analyzed (Participants) | 1 | 1
  Participant 3, PET Scan 3, Day 4 | 2.77 | 2.62
  Participant 4, PET Scan 1, Baseline: number analyzed (Participants) | 1 | 1
  Participant 4, PET Scan 1, Baseline | 13.62 | 14.90
  Participant 4, PET Scan 2, Day 1: number analyzed (Participants) | 1 | 1
  Participant 4, PET Scan 2, Day 1 | 2.07 | 2.11
  Participant 4, PET Scan 3, Day 4: number analyzed (Participants) | 1 | 0
  Participant 4, PET Scan 3, Day 4 | 2.84 |
  Participant 4, PET Scan 3, Day 10: number analyzed (Participants) | 0 | 1
  Participant 4, PET Scan 3, Day 10 |  | 7.72

3. Primary Outcome: Regional VT of [18F]-IMA601 in Anterior Cingulate at Each Brain Scan
Description: Regional VT of [18F]-IMA601 in anterior cingulate at each brain scan was measured with a PET scan. Participants received an IV dose of the radiolabelled tracer, [18F]-IMA601, at the start of each PET scan. Participant wise data was reported for this outcome measure.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Number; unit: mL/cm^3
Arm/Group | Group 1: ASN51 Low Dose | Group 2: ASN51 High Dose
Number analyzed (Participants) | 4 | 4
mL/cm^3
  Participant 1, PET Scan 1, Baseline: number analyzed (Participants) | 1 | 1
  Participant 1, PET Scan 1, Baseline | 13.57 | 18.51
  Participant 1, PET Scan 2, Day 1: number analyzed (Participants) | 1 | 1
  Participant 1, PET Scan 2, Day 1 | 1.97 | 1.60
  Participant 1, PET Scan 3, Day 4: number analyzed (Participants) | 1 | 1
  Participant 1, PET Scan 3, Day 4 | 2.85 | 3.98
  Participant 2, PET Scan 1, Baseline: number analyzed (Participants) | 1 | 1
  Participant 2, PET Scan 1, Baseline | 17.45 | 16.08
  Participant 2, PET Scan 2, Day 1: number analyzed (Participants) | 1 | 1
  Participant 2, PET Scan 2, Day 1 | 2.13 | 2.56
  Participant 2, PET Scan 3, Day 4: number analyzed (Participants) | 0 | 1
  Participant 2, PET Scan 3, Day 4 |  | 3.17
  Participant 2, PET Scan 3, Day 9: number analyzed (Participants) | 1 | 0
  Participant 2, PET Scan 3, Day 9 | 19.79 |
  Participant 3, PET Scan 1, Baseline: number analyzed (Participants) | 1 | 1
  Participant 3, PET Scan 1, Baseline | 18.34 | 20.14
  Participant 3, PET Scan 2, Day 1: number analyzed (Participants) | 1 | 1
  Participant 3, PET Scan 2, Day 1 | 2.26 | 1.60
  Participant 3, PET Scan 3, Day 4: number analyzed (Participants) | 1 | 1
  Participant 3, PET Scan 3, Day 4 | 2.94 | 2.82
  Participant 4, PET Scan 1, Baseline: number analyzed (Participants) | 1 | 1
  Participant 4, PET Scan 1, Baseline | 15.87 | 17.02
  Participant 4, PET Scan 2, Day 1: number analyzed (Participants) | 1 | 1
  Participant 4, PET Scan 2, Day 1 | 1.94 | 2.04
  Participant 4, PET Scan 3, Day 4: number analyzed (Participants) | 1 | 0
  Participant 4, PET Scan 3, Day 4 | 2.69 |
  Participant 4, PET Scan 3, Day 10: number analyzed (Participants) | 0 | 1
  Participant 4, PET Scan 3, Day 10 |  | 8.53

4. Primary Outcome: Regional VT of [18F]-IMA601 in Caudate at Each Brain Scan
Description: Regional VT of [18F]-IMA601 in Caudate at each brain scan was measured with a PET scan. Participants received an IV dose of the radiolabelled tracer, [18F]-IMA601, at the start of each PET scan. Participant wise data was reported for this outcome measure.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Number; unit: mL/cm^3
Arm/Group | Group 1: ASN51 Low Dose | Group 2: ASN51 High Dose
Number analyzed (Participants) | 4 | 4
mL/cm^3
  Participant 1, PET Scan 1, Baseline: number analyzed (Participants) | 1 | 1
  Participant 1, PET Scan 1, Baseline | 8.25 | 13.28
  Participant 1, PET Scan 2, Day 1: number analyzed (Participants) | 1 | 1
  Participant 1, PET Scan 2, Day 1 | 1.21 | 1.23
  Participant 1, PET Scan 3, Day 4: number analyzed (Participants) | 1 | 1
  Participant 1, PET Scan 3, Day 4 | 1.76 | 2.97
  Participant 2, PET Scan 1, Baseline: number analyzed (Participants) | 1 | 1
  Participant 2, PET Scan 1, Baseline | 12.89 | 11.43
  Participant 2, PET Scan 2, Day 1: number analyzed (Participants) | 1 | 1
  Participant 2, PET Scan 2, Day 1 | 1.74 | 2.32
  Participant 2, PET Scan 3, Day 4: number analyzed (Participants) | 0 | 1
  Participant 2, PET Scan 3, Day 4 |  | 2.75
  Participant 2, PET Scan 3, Day 9: number analyzed (Participants) | 1 | 0
  Participant 2, PET Scan 3, Day 9 | 14.98 |
  Participant 3, PET Scan 1, Baseline: number analyzed (Participants) | 1 | 1
  Participant 3, PET Scan 1, Baseline | 13.77 | 13.95
  Participant 3, PET Scan 2, Day 1: number analyzed (Participants) | 1 | 1
  Participant 3, PET Scan 2, Day 1 | 1.77 | 1.17
  Participant 3, PET Scan 3, Day 4: number analyzed (Participants) | 1 | 1
  Participant 3, PET Scan 3, Day 4 | 2.27 | 1.94
  Participant 4, PET Scan 1, Baseline: number analyzed (Participants) | 1 | 1
  Participant 4, PET Scan 1, Baseline | 11.50 | 13.44
  Participant 4, PET Scan 2, Day 1: number analyzed (Participants) | 1 | 1
  Participant 4, PET Scan 2, Day 1 | 1.66 | 1.91
  Participant 4, PET Scan 3, Day 4: number analyzed (Participants) | 1 | 0
  Participant 4, PET Scan 3, Day 4 | 2.04 |
  Participant 4, PET Scan 3, Day 10: number analyzed (Participants) | 0 | 1
  Participant 4, PET Scan 3, Day 10 |  | 6.99

5. Primary Outcome: Regional VT of [18F]-IMA601 in Putamen at Each Brain Scan
Description: Regional VT of [18F]-IMA601 in Putamen at each brain scan was measured with a PET scan. Participants received an IV dose of the radiolabelled tracer, [18F]-IMA601, at the start of each PET scan.
  Participant wise data was reported for this outcome measure.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Number; unit: mL/cm^3
Arm/Group | Group 1: ASN51 Low Dose | Group 2: ASN51 High Dose
Number analyzed (Participants) | 4 | 4
mL/cm^3
  Participant 1, PET Scan 1, Baseline: number analyzed (Participants) | 1 | 1
  Participant 1, PET Scan 1, Baseline | 12.74 | 17.00
  Participant 1, PET Scan 2, Day 1: number analyzed (Participants) | 1 | 1
  Participant 1, PET Scan 2, Day 1 | 2.03 | 1.63
  Participant 1, PET Scan 3, Day 4: number analyzed (Participants) | 1 | 1
  Participant 1, PET Scan 3, Day 4 | 2.86 | 3.89
  Participant 2, PET Scan 1, Baseline: number analyzed (Participants) | 1 | 1
  Participant 2, PET Scan 1, Baseline | 17.46 | 15.89
  Participant 2, PET Scan 2, Day 1: number analyzed (Participants) | 1 | 1
  Participant 2, PET Scan 2, Day 1 | 2.32 | 2.76
  Participant 2, PET Scan 3, Day 4: number analyzed (Participants) | 0 | 1
  Participant 2, PET Scan 3, Day 4 |  | 3.35
  Participant 2, PET Scan 3, Day 9: number analyzed (Participants) | 1 | 0
  Participant 2, PET Scan 3, Day 9 | 20.27 |
  Participant 3, PET Scan 1, Baseline: number analyzed (Participants) | 1 | 1
  Participant 3, PET Scan 1, Baseline | 16.76 | 20.70
  Participant 3, PET Scan 2, Day 1: number analyzed (Participants) | 1 | 1
  Participant 3, PET Scan 2, Day 1 | 2.31 | 1.78
  Participant 3, PET Scan 3, Day 4: number analyzed (Participants) | 1 | 1
  Participant 3, PET Scan 3, Day 4 | 2.87 | 2.96
  Participant 4, PET Scan 1, Baseline: number analyzed (Participants) | 1 | 1
  Participant 4, PET Scan 1, Baseline | 14.88 | 17.00
  Participant 4, PET Scan 2, Day 1: number analyzed (Participants) | 1 | 1
  Participant 4, PET Scan 2, Day 1 | 2.02 | 2.07
  Participant 4, PET Scan 3, Day 4: number analyzed (Participants) | 1 | 0
  Participant 4, PET Scan 3, Day 4 | 2.74 |
  Participant 4, PET Scan 3, Day 10: number analyzed (Participants) | 0 | 1
  Participant 4, PET Scan 3, Day 10 |  | 8.50

6. Primary Outcome: Regional VT of [18F]-IMA601 in Accumbens at Each Brain Scan
Description: Regional VT of [18F]-IMA601 in Accumbens at each brain scan was measured with a PET scan. Participants received an IV dose of the radiolabelled tracer, [18F]-IMA601, at the start of each PET scan. Participant wise data was reported for this outcome measure.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Number; unit: mL/cm^3
Arm/Group | Group 1: ASN51 Low Dose | Group 2: ASN51 High Dose
Number analyzed (Participants) | 4 | 4
mL/cm^3
  Participant 1, PET Scan 1, Baseline: number analyzed (Participants) | 1 | 1
  Participant 1, PET Scan 1, Baseline | 13.16 | 19.29
  Participant 1, PET Scan 2, Day 1: number analyzed (Participants) | 1 | 1
  Participant 1, PET Scan 2, Day 1 | 1.73 | 1.51
  Participant 1, PET Scan 3, Day 4: number analyzed (Participants) | 1 | 1
  Participant 1, PET Scan 3, Day 4 | 2.51 | 3.91
  Participant 2, PET Scan 1, Baseline: number analyzed (Participants) | 1 | 1
  Participant 2, PET Scan 1, Baseline | 18.94 | 16.58
  Participant 2, PET Scan 2, Day 1: number analyzed (Participants) | 1 | 1
  Participant 2, PET Scan 2, Day 1 | 2.22 | 2.66
  Participant 2, PET Scan 3, Day 4: number analyzed (Participants) | 0 | 1
  Participant 2, PET Scan 3, Day 4 |  | 3.29
  Participant 2, PET Scan 3, Day 9: number analyzed (Participants) | 1 | 0
  Participant 2, PET Scan 3, Day 9 | 22.18 |
  Participant 3, PET Scan 1, Baseline: number analyzed (Participants) | 1 | 1
  Participant 3, PET Scan 1, Baseline | 18.57 | 20.52
  Participant 3, PET Scan 2, Day 1: number analyzed (Participants) | 1 | 1
  Participant 3, PET Scan 2, Day 1 | 2.14 | 1.49
  Participant 3, PET Scan 3, Day 4: number analyzed (Participants) | 1 | 1
  Participant 3, PET Scan 3, Day 4 | 2.80 | 2.67
  Participant 4, PET Scan 1, Baseline: number analyzed (Participants) | 1 | 1
  Participant 4, PET Scan 1, Baseline | 16.18 | 18.65
  Participant 4, PET Scan 2, Day 1: number analyzed (Participants) | 1 | 1
  Participant 4, PET Scan 2, Day 1 | 1.87 | 2.64
  Participant 4, PET Scan 3, Day 4: number analyzed (Participants) | 1 | 0
  Participant 4, PET Scan 3, Day 4 | 2.62 |
  Participant 4, PET Scan 3, Day 10: number analyzed (Participants) | 0 | 1
  Participant 4, PET Scan 3, Day 10 |  | 9.09

7. Primary Outcome: Regional VT of [18F]-IMA601 in Amygdala at Each Brain Scan
Description: Regional VT of [18F]-IMA601 in Amygdala at each brain scan was measured with a PET scan. Participants received an IV dose of the radiolabelled tracer, [18F]-IMA601, at the start of each PET scan. Participant wise data was reported for this outcome measure.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Number; unit: mL/cm^3
Arm/Group | Group 1: ASN51 Low Dose | Group 2: ASN51 High Dose
Number analyzed (Participants) | 4 | 4
mL/cm^3
  Participant 1, PET Scan 1, Baseline: number analyzed (Participants) | 1 | 1
  Participant 1, PET Scan 1, Baseline | 15.00 | 18.91
  Participant 1, PET Scan 2, Day 1: number analyzed (Participants) | 1 | 1
  Participant 1, PET Scan 2, Day 1 | 2.13 | 1.54
  Participant 1, PET Scan 3, Day 4: number analyzed (Participants) | 1 | 1
  Participant 1, PET Scan 3, Day 4 | 3.13 | 4.42
  Participant 2, PET Scan 1, Baseline: number analyzed (Participants) | 1 | 1
  Participant 2, PET Scan 1, Baseline | 19.84 | 17.77
  Participant 2, PET Scan 2, Day 1: number analyzed (Participants) | 1 | 1
  Participant 2, PET Scan 2, Day 1 | 2.30 | 2.50
  Participant 2, PET Scan 3, Day 4: number analyzed (Participants) | 0 | 1
  Participant 2, PET Scan 3, Day 4 |  | 3.40
  Participant 2, PET Scan 3, Day 9: number analyzed (Participants) | 1 | 0
  Participant 2, PET Scan 3, Day 9 | 22.25 |
  Participant 3, PET Scan 1, Baseline: number analyzed (Participants) | 1 | 1
  Participant 3, PET Scan 1, Baseline | 19.37 | 22.00
  Participant 3, PET Scan 2, Day 1: number analyzed (Participants) | 1 | 1
  Participant 3, PET Scan 2, Day 1 | 2.32 | 1.76
  Participant 3, PET Scan 3, Day 4: number analyzed (Participants) | 1 | 1
  Participant 3, PET Scan 3, Day 4 | 3.11 | 3.12
  Participant 4, PET Scan 1, Baseline: number analyzed (Participants) | 1 | 1
  Participant 4, PET Scan 1, Baseline | 16.77 | 17.57
  Participant 4, PET Scan 2, Day 1: number analyzed (Participants) | 1 | 1
  Participant 4, PET Scan 2, Day 1 | 1.89 | 2.10
  Participant 4, PET Scan 3, Day 4: number analyzed (Participants) | 1 | 0
  Participant 4, PET Scan 3, Day 4 | 2.94 |
  Participant 4, PET Scan 3, Day 10: number analyzed (Participants) | 0 | 1
  Participant 4, PET Scan 3, Day 10 |  | 9.38

8. Primary Outcome: Regional VT of [18F]-IMA601 in Cerebral White Matter at Each Brain Scan
Description: Regional VT of [18F]-IMA601 in cerebral white matter at each brain scan was measured with a PET scan. Participants received an IV dose of the radiolabelled tracer, [18F]-IMA601, at the start of each PET scan. Participant wise data was reported for this outcome measure.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Number; unit: mL/cm^3
Arm/Group | Group 1: ASN51 Low Dose | Group 2: ASN51 High Dose
Number analyzed (Participants) | 4 | 4
mL/cm^3
  Participant 1, PET Scan 1, Baseline: number analyzed (Participants) | 1 | 1
  Participant 1, PET Scan 1, Baseline | 8.39 | 10.72
  Participant 1, PET Scan 2, Day 1: number analyzed (Participants) | 1 | 1
  Participant 1, PET Scan 2, Day 1 | 1.67 | 1.32
  Participant 1, PET Scan 3, Day 4: number analyzed (Participants) | 1 | 1
  Participant 1, PET Scan 3, Day 4 | 2.30 | 2.96
  Participant 2, PET Scan 1, Baseline: number analyzed (Participants) | 1 | 1
  Participant 2, PET Scan 1, Baseline | 11.39 | 10.15
  Participant 2, PET Scan 2, Day 1: number analyzed (Participants) | 1 | 1
  Participant 2, PET Scan 2, Day 1 | 1.89 | 2.43
  Participant 2, PET Scan 3, Day 4: number analyzed (Participants) | 0 | 1
  Participant 2, PET Scan 3, Day 4 |  | 2.96
  Participant 2, PET Scan 3, Day 9: number analyzed (Participants) | 1 | 0
  Participant 2, PET Scan 3, Day 9 | 13.25 |
  Participant 3, PET Scan 1, Baseline: number analyzed (Participants) | 1 | 1
  Participant 3, PET Scan 1, Baseline | 12.39 | 12.86
  Participant 3, PET Scan 2, Day 1: number analyzed (Participants) | 1 | 1
  Participant 3, PET Scan 2, Day 1 | 2.03 | 1.51
  Participant 3, PET Scan 3, Day 4: number analyzed (Participants) | 1 | 1
  Participant 3, PET Scan 3, Day 4 | 2.46 | 2.45
  Participant 4, PET Scan 1, Baseline: number analyzed (Participants) | 1 | 1
  Participant 4, PET Scan 1, Baseline | 9.95 | 11.45
  Participant 4, PET Scan 2, Day 1: number analyzed (Participants) | 1 | 1
  Participant 4, PET Scan 2, Day 1 | 1.81 | 1.78
  Participant 4, PET Scan 3, Day 4: number analyzed (Participants) | 1 | 0
  Participant 4, PET Scan 3, Day 4 | 2.34 |
  Participant 4, PET Scan 3, Day 10: number analyzed (Participants) | 0 | 1
  Participant 4, PET Scan 3, Day 10 |  | 6.34

9. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious TEAEs
Description: An adverse event (AE) is defined as any untoward medical occurrence in a participant or clinical trial subject administered a medicinal product and which does not necessarily have a causal relationship with that treatment. A TEAE is defined as an AE that emerges during treatment (having been absent before treatment) or that worsens after treatment. Serious TEAE is defined as any adverse event that is fatal, is life-threatening, requires or prolongs in-patient treatment, results in persistent or significant disability or incapacity, or is a congenital anomaly or birth defect.
Time Frame: Up to 4.5 months
Population: Safety population included all participants who received at least one dose of the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: ASN51 Low Dose | Group 2: ASN51 High Dose
Number analyzed (Participants) | 6 | 6
Participants
  Participants with TEAEs | 4 | 3
  Participants with Serious TEAEs | 0 | 0

10. Secondary Outcome: Number of Participants With Clinically Significant Abnormalities in Vital Signs
Description: Vital signs including blood pressure, pulse rate, tympanic temperature, and respiratory rate were assessed. Number of participants with clinically significant abnormalities in vital signs were reported. Clinical significance was determined by the investigator.
Time Frame: Up to 4.5 months
Population: Safety population included participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: ASN51 Low Dose | Group 2: ASN51 High Dose
Number analyzed (Participants) | 6 | 6
Participants | 0 | 0

11. Secondary Outcome: Number of Participants With Clinically Significant Abnormal 12-lead Safety Electrocardiogram (ECG) Findings
Description: ECG parameters including Ventricular rate, QRS complex of the ECG reflects the rapid depolarization of the right and left ventricles (QRS) interval, portion of the ECG between consecutive R waves, representing the ventricular rate (PR) interval, and QTc interval with Fridericia's correction method (QTcF) was measured. Number of participants with clinically significant abnormal ECG findings were reported. Clinical significance was determined by the investigator.
Time Frame: Up to 4.5 months
Population: Safety population included participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: ASN51 Low Dose | Group 2: ASN51 High Dose
Number analyzed (Participants) | 6 | 6
Participants | 0 | 0

12. Secondary Outcome: Number of Participants With Clinically Significant Abnormal Physical Examinations
Description: Complete physical examination including general appearance; head, ears, eyes, nose and throat; thyroid; lymph nodes; back and neck; heart; chest; lungs; abdomen; skin; and extremities were performed. Number of participants with clinically significant abnormal physical examinations were reported. Clinical significance was determined by the investigator.
Time Frame: Up to 4.5 months
Population: Safety population included participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: ASN51 Low Dose | Group 2: ASN51 High Dose
Number analyzed (Participants) | 6 | 6
Participants | 0 | 0

13. Secondary Outcome: Number of Participants With Clinically Significant Abnormal Neurological Examinations Findings
Description: Complete neurological examinations including motor system, romberg test, coordination, and direct pupillary reflexes were performed. Number of participants with clinically significant abnormal neurological examinations findings were reported. Clinical significance was determined by the investigator.
Time Frame: Up to 4.5 months
Population: Safety population included participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: ASN51 Low Dose | Group 2: ASN51 High Dose
Number analyzed (Participants) | 6 | 6
Participants | 0 | 0

14. Secondary Outcome: Number of Participants With Clinically Significant Changes in Laboratory Parameters
Description: Laboratory tests including hematology, clinical chemistry, coagulation, serology, follicle stimulating hormone (FSH) test (only for females), and urinalysis were performed. Number of participants with clinically significant changes in laboratory parameters were reported. Clinical significance was determined by the investigator.
Time Frame: Up to 4.5 months
Population: Safety population included participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: ASN51 Low Dose | Group 2: ASN51 High Dose
Number analyzed (Participants) | 6 | 6
Participants | 0 | 0

15. Secondary Outcome: Number of Participants With Suicidal Ideation According to Columbia - Suicide Severity Rating Scale (C-SSRS) Ideation
Description: The C-SSRS is a valid and reliable suicidal scale that includes a seven-item subscale that asks participants to self-report on actual attempts, interrupted attempts, aborted attempts, and preparatory acts or behaviors. The suicidal ideation section is rated on a scale from 1 to 5, with higher score indicating a greater severity of suicidal ideation or risk of suicidal behavior. Participants who respond "yes" to any question related to suicidal ideation are reported in this outcome measure.
Time Frame: Up to 4.5 months
Population: Safety population included participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: ASN51 Low Dose | Group 2: ASN51 High Dose
Number analyzed (Participants) | 6 | 6
Participants | 0 | 0

16. Secondary Outcome: Plasma Concentration of ASN51 at Each Post-dose PET Scan
Time Frame: Day 1: 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 16 hours; Day 11: 8 hours; Day 14: 0.25, 0.5, 1, 2, 4, 6, 12 hours; Day 15, Day 16, Day 17, Day 18, Day 20, and Day 23
Population: PK analysis population included the participants who provided evaluable data for the comparisons of interest. These participants had at least one quantifiable plasma concentration. Number analyzed is the number of participants with data available for analysis at a specified time point.
Measure: Mean (Standard Deviation); unit: nanograms/milliliter (ng/mL)
Arm/Group | Group 1: ASN51 Low Dose | Group 2: ASN51 High Dose
Number analyzed (Participants) | 6 | 6
nanograms/milliliter (ng/mL)
  Day 1: 0.25 hour post-dose: number analyzed (Participants) | 5 | 4
  Day 1: 0.25 hour post-dose | 4.833 (11.839) | 20.18 (31.680)
  Day 1: 0.5 hour post-dose | 132.9 (65.354) | 232.7 (228.23)
  Day 1: 1 hour post-dose | 173.8 (28.174) | 355.3 (66.704)
  Day 1: 1.5 hours post-dose: number analyzed (Participants) | 5 | 4
  Day 1: 1.5 hours post-dose | 155.2 (11.089) | 311.3 (40.934)
  Day 1: 2 hours post-dose: number analyzed (Participants) | 6 | 4
  Day 1: 2 hours post-dose | 152.5 (13.867) | 310.3 (45.559)
  Day 1: 3 hours post-dose: number analyzed (Participants) | 5 | 6
  Day 1: 3 hours post-dose | 155.2 (11.476) | 277.3 (40.143)
  Day 1: 4 hours post-dose | 140.3 (21.630) | 281.8 (34.032)
  Day 1: 6 hours post-dose | 125.7 (11.183) | 254.7 (38.568)
  Day 1: 8 hours post-dose | 123.8 (7.2503) | 244.0 (28.071)
  Day 1: 12 hours post-dose | 97.30 (8.8050) | 199.2 (31.212)
  Day 1: 16 hours post-dose | 82.98 (4.2687) | 154.3 (23.036)
  Day 11: 8 hours post-dose | 326.0 (43.253) | 567.3 (228.33)
  Day 14: 0.25 hour post-dose | 264.2 (55.333) | 416.2 (175.02)
  Day 14: 0.5 hour post-dose | 417.8 (130.39) | 541.7 (224.05)
  Day 14: 1 hour post-dose | 427.8 (54.455) | 682.5 (280.47)
  Day 14: 2 hours post-dose | 398.8 (46.525) | 695.3 (285.19)
  Day 14: 4 hours post-dose | 362.2 (46.357) | 640.2 (258.28)
  Day 14: 6 hours post-dose | 339.2 (28.117) | 599.0 (255.59)
  Day 14: 12 hours post-dose | 268.0 (28.390) | 499.2 (214.34)
  Day 15 | 242.3 (33.279) | 455.8 (180.41)
  Day 16 | 150.2 (26.347) | 295.4 (134.63)
  Day 17: number analyzed (Participants) | 3 | 3
  Day 17 | 97.23 (17.151) | 105.8 (40.751)
  Day 18 | 63.52 (22.281) | 141.0 (69.510)
  Day 20 | 29.38 (15.536) | 78.52 (45.813)
  Day 23: number analyzed (Participants) | 1 | 6
  Day 23 | 11.01 (11.685) | 35.24 (33.575)

17. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of ASN51
Description: Cmax was obtained directly from the concentration-time data.
Time Frame: Pre-dose, and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 16 hours post-dose on Day 1; Pre-dose, and 0.25, 0.5, 1, 2, 4, 6, and 12 hours post-dose on Day 14
Population: PK analysis population included participants who had evaluable data for the comparisons of interest. These participants had at least one quantifiable plasma concentration.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Group 1: ASN51 Low Dose | Group 2: ASN51 High Dose
Number analyzed (Participants) | 6 | 6
ng/mL
  Day 1 | 183 (14.8) | 386 (30.4)
  Day 14 | 462 (20.0) | 624 (71.8)

18. Secondary Outcome: Dose-normalised Cmax (Cmax/Dose) of ASN51
Description: Calculated as Cmax /Dose administered.
Time Frame: Pre-dose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 16 hours post-dose on Day 1; Pre-dose and 0.25, 0.5, 1, 2, 4, 6, and 12 hours post-dose on Day 14
Population: as for outcome 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL/milligram (mg)
Arm/Group | Group 1: ASN51 Low Dose | Group 2: ASN51 High Dose
Number analyzed (Participants) | 6 | 6
ng/mL/milligram (mg)
  Day 1 | 18.3 (14.8) | 19.3 (30.4)
  Day 14 | 46.2 (20.0) | 31.2 (71.8)

19. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of ASN51
Description: The tmax was obtained directly from the concentration-time data.
Time Frame: as for outcome 18
Population: as for outcome 17
Measure: Median (Full Range); unit: hours
Arm/Group | Group 1: ASN51 Low Dose | Group 2: ASN51 High Dose
Number analyzed (Participants) | 6 | 6
hours
  Day 1 | 1.00 [0.500 to 1.50] | 1.00 [0.500 to 2.05]
  Day 14 | 0.767 [0.500 to 2.00] | 2.00 [1.00 to 2.00]

20. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to Infinity (AUCinf) of ASN51
Description: AUCinf was calculated using the trapezoidal method for the interval 0 to tlast (time tlast is the time at which the last non-zero level was recorded), plus the area under the exponential curve from tlast to infinity.
Time Frame: Pre-dose and 0.25, 0.5, 1, 2, 4, 6, and 12 hours post-dose on Day 14
Population: as for outcome 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*nanograms/milliliters (h*ng/mL)
Arm/Group | Group 1: ASN51 Low Dose | Group 2: ASN51 High Dose
Number analyzed (Participants) | 6 | 6
hours*nanograms/milliliters (h*ng/mL) | 20428 (24.3) | 40365 (56.3)

21. Secondary Outcome: Dose-normalised AUC Infinity (AUCinf /D) of ASN51
Description: Calculated as AUCinf /Dose administered. Here, the unit of measure is represented as hours*nanograms per milliliters per milligram (h*ng/mL/mg).
Time Frame: Pre-dose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 16 hours post-dose on Day 1, Pre-dose and 0.25, 0.5, 1, 2, 4, 6, and 12 hours post-dose on Day 14
Population: as for outcome 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL/mg
Arm/Group | Group 1: ASN51 Low Dose | Group 2: ASN51 High Dose
Number analyzed (Participants) | 6 | 6
h*ng/mL/mg | 2043 (24.3) | 2018 (56.3)

22. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to Time of Last Measurable Concentration (AUClast) of ASN51
Description: AUClast was calculated using the trapezoidal method.
Time Frame: Pre-dose and 0.25, 0.5, 1, 2, 4, 6, and 12 hours post-dose on Day 14
Population: as for outcome 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Group 1: ASN51 Low Dose | Group 2: ASN51 High Dose
Number analyzed (Participants) | 6 | 6
h*ng/mL | 19655 (21.3) | 36574 (60.6)

23. Secondary Outcome: Area Under the Plasma Concentration-time Curve During a Dosing Interval (AUCtau) of ASN51
Description: AUCtau was calculated using the trapezoidal method.
Time Frame: as for outcome 21
Population: as for outcome 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Group 1: ASN51 Low Dose | Group 2: ASN51 High Dose
Number analyzed (Participants) | 6 | 6
h*ng/mL
  Day 1 | 2527 (8.2) | 4888 (15.1)
  Day 14 | 7067 (11.6) | 11237 (73.4)

24. Secondary Outcome: Terminal Half-life (t1/2) of ASN51
Description: The t1/2 was calculated from the terminal slope of the log concentration-time curve as follows: t1/2 = loge 2 / lambda(λ)z.
Time Frame: Pre-dose and 0.25, 0.5, 1, 2, 4, 6, and 12 hours post-dose on Day 14
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Group 1: ASN51 Low Dose | Group 2: ASN51 High Dose
Number analyzed (Participants) | 6 | 6
hours | 45.1 (13.9) | 66.0 (25.8)

25. Secondary Outcome: Terminal Rate Constant (λz) of ASN51
Description: Terminal rate constant was estimated by linear regression of logarithmically transformed concentration versus time data.
Time Frame: Pre-dose and 0.25, 0.5, 1, 2, 4, 6, and 12 hours post-dose on Day 14
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: 1 per hour (1/h)
Arm/Group | Group 1: ASN51 Low Dose | Group 2: ASN51 High Dose
Number analyzed (Participants) | 6 | 6
1 per hour (1/h) | 0.0163 (0.00392) | 0.0119 (0.00444)

26. Secondary Outcome: Apparent Total Clearance From Plasma After Oral Administration (CLss/F) of ASN51 at Steady State
Description: Calculated using the formula as follows: CLss/F = Dose/ AUCtau.
Time Frame: Pre-dose and 0.25, 0.5, 1, 2, 4, 6, and 12 hours post-dose on Day 14
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Liters/hour (L/h)
Arm/Group | Group 1: ASN51 Low Dose | Group 2: ASN51 High Dose
Number analyzed (Participants) | 6 | 6
Liters/hour (L/h) | 1.42 (0.174) | 2.25 (2.12)

27. Secondary Outcome: Apparent Volume of Distribution After Oral Administration (VZ/F) of ASN51
Description: Calculated using the formula as follows: VZ/F = Dose/λz *AUCtau.
Time Frame: Pre-dose, 0.25, 0.5, 1, 2, 4, 6, and 12 hours post-dose on Day 14
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Group 1: ASN51 Low Dose | Group 2: ASN51 High Dose
Number analyzed (Participants) | 6 | 6
Liters | 92.1 (28.9) | 254 (340)

28. Secondary Outcome: Trough Plasma Concentration (Ctrough) of ASN51
Description: Trough plasma concentration i.e., measured concentration at the end of a dosing interval at steady state (taken directly before next administration, and at 1 dosing interval after the final dose) was obtained directly from the concentration-time data.
Time Frame: Pre-dose on Days 2, 4, 7, 11 and 14; and 8 hours post-dose on Day 11; 0.25, 0.5, 1, 2, 4, 6, and 12 hours post-dose on Day 14, and on Day 15
Population: as for outcome 17
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Group 1: ASN51 Low Dose | Group 2: ASN51 High Dose
Number analyzed (Participants) | 6 | 6
ng/mL
  Day 2 | 82.4 [71.3 to 95.2] | 149 [112 to 180]
  Day 4 | 173 [148 to 201] | 316 [247 to 404]
  Day 7 | 227 [195 to 263] | 444 [365 to 539]
  Day 11 | 238 [202 to 279] | 431 [284 to 654]
  Day 14 | 236 [199 to 280] | 377 [179 to 795]
  Day 15 | 240 [206 to 281] | 405 [210 to 778]

29. Secondary Outcome: Accumulation Ratio for AUC (Rac[AUC]) of ASN51
Description: Accumulation ratio was calculated from area under the plasma concentration-time curve during a dosing interval at steady state, and after single dose of ASN51.
Time Frame: Pre-dose up to Day 14
Population: as for outcome 17
Measure: Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Group 1: ASN51 Low Dose | Group 2: ASN51 High Dose
Number analyzed (Participants) | 6 | 6
Ratio | 2.81 [2.52 to 3.09] | 2.52 [1.60 to 3.44]

30. Secondary Outcome: Accumulation Ratio for Cmax (Rac[Cmax]) of ASN51
Description: Rac(Cmax) was calculated from Cmax at steady state and Cmax after single dose.
Time Frame: Pre-dose up to Day 14
Population: as for outcome 17
Measure: Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Group 1: ASN51 Low Dose | Group 2: ASN51 High Dose
Number analyzed (Participants) | 6 | 6
Ratio | 2.55 [2.22 to 2.88] | 1.74 [1.12 to 2.37]

31. Secondary Outcome: Effect of Food on PBMC Protein O-GlcNAcylation Levels During Repeated Dosing of ASN51
Description: The analysis of the PD response of PBMCs during repeated ASN51 dosing was conducted using ANOVA. Assessments were conducted at pre-dose and 8 hours post-dose on Day 11 (fed state) and Day 14 (fasted state). The ratio of fed to fasted has been reported.
Time Frame: Predose and 8 hours post-dose on Days 11 and 14
Population: PD analysis population included all participants in the safety population for who a PBMC measure is available.
Measure: Geometric Mean (90% Confidence Interval); unit: Ratios
Arm/Group | Group 1: ASN51 Low Dose | Group 2: ASN51 High Dose
Number analyzed (Participants) | 6 | 6
Ratios
  Predose | 0.87 [0.56 to 1.35] | 1.05 [0.56 to 1.97]
  8 hours post-dose | 0.94 [0.69 to 1.28] | 0.86 [0.55 to 1.34]

32. Secondary Outcome: Group 1: Estimated O-GlcNAcase Receptor Occupancy (RO) by Plasma Concentration of ASN51 and Time
Description: Occupancy estimates were plotted against plasma concentrations of ASN51, corresponding to the start of each post-dose PET scan. Participant wise data was reported for this outcome measure.
  Row titles include participant number, PET scan session, post-dose time, and plasma concentration.
Time Frame: At 5.1, 75.9 hours post-dose on Day 1 (Participant 1); 6.0, 196.9 hours post-dose on Day 1 (Participant 2); 5.2, 79.3 hours post-dose on Day 1 (Participant 3) and 5.5 and 77.0 hours post-dose on Day 1 (Participant 4)
Population: PET population included all participants in the safety population who had a baseline PET scan, at least 1 post-baseline PET scan, and a PK result immediately preceding a PET scan. No summary analysis was done due to low number of participants, therefore participant wise data are reported.
Measure: Number; unit: percentage of receptor occupancy
Arm/Group | Group 1: ASN51 Low Dose
Number analyzed (Participants) | 4
percentage of receptor occupancy
  Participant 1: PET Scan 2, 5.1 hours at 118.0 ng/mL: number analyzed (Participants) | 1
  Participant 1: PET Scan 2, 5.1 hours at 118.0 ng/mL | 92.0
  Participant 1: PET Scan 3, 75.9 hours at 101.0 ng/mL: number analyzed (Participants) | 1
  Participant 1: PET Scan 3, 75.9 hours at 101.0 ng/mL | 84.6
  Participant 2: PET Scan 2, 6.0 hours at 118.0 ng/mL: number analyzed (Participants) | 1
  Participant 2: PET Scan 2, 6.0 hours at 118.0 ng/mL | 94.3
  Participant 2: PET Scan 3, 196.9 hours at 4.8 ng/mL: number analyzed (Participants) | 1
  Participant 2: PET Scan 3, 196.9 hours at 4.8 ng/mL | -16.0
  Participant 3: PET Scan 2, 5.2 hours at 121.0 ng/mL: number analyzed (Participants) | 1
  Participant 3: PET Scan 2, 5.2 hours at 121.0 ng/mL | 95.6
  Participant 3: PET Scan 3, 79.3 hours at 127.0 ng/mL: number analyzed (Participants) | 1
  Participant 3: PET Scan 3, 79.3 hours at 127.0 ng/mL | 91.3
  Participant 4: PET Scan 2, 5.5 hours at 171.0 ng/mL: number analyzed (Participants) | 1
  Participant 4: PET Scan 2, 5.5 hours at 171.0 ng/mL | 97.8
  Participant 4: PET Scan 3, 77.0 hours at 91.4 ng/mL: number analyzed (Participants) | 1
  Participant 4: PET Scan 3, 77.0 hours at 91.4 ng/mL | 91.9

33. Secondary Outcome: Group 2: Estimated O-GlcNAcase RO by Plasma Concentration of ASN51 and Time
Description: as for outcome 32
Time Frame: At 5.5, 75.6 hours post-dose on Day 1 (Participant 5); 5.3, 75.4 hours post-dose on Day 1 (Participant 6); 4.9, 75.9 hours post-dose on Day 1 (Participant 7) and 5.0 and 220.5 hours post-dose on Day 1 (Participant 8)
Population: as for outcome 32
Measure: Number; unit: percentage of receptor occupancy
Arm/Group | Group 2: ASN51 High Dose
Number analyzed (Participants) | 4
percentage of receptor occupancy
  Participant 5: PET Scan 2, 5.5 hours at 232.0 ng/mL: number analyzed (Participants) | 1
  Participant 5: PET Scan 2, 5.5 hours at 232.0 ng/mL | 98.5
  Participant 5: PET Scan 3, 75.6 hours at 67.3 ng/mL: number analyzed (Participants) | 1
  Participant 5: PET Scan 3, 75.6 hours at 67.3 ng/mL | 83.4
  Participant 6: PET Scan 2, 5.3 hours at 309.0 ng/mL: number analyzed (Participants) | 1
  Participant 6: PET Scan 2, 5.3 hours at 309.0 ng/mL | 98.1
  Participant 6: PET Scan 3, 75.4 hours at 152.0 ng/mL: number analyzed (Participants) | 1
  Participant 6: PET Scan 3, 75.4 hours at 152.0 ng/mL | 93.3
  Participant 7: PET Scan 2, 4.9 hours at 267.0 ng/mL: number analyzed (Participants) | 1
  Participant 7: PET Scan 2, 4.9 hours at 267.0 ng/mL | 98.1
  Participant 7: PET Scan 3, 75.9 hours at 132.0 ng/mL: number analyzed (Participants) | 1
  Participant 7: PET Scan 3, 75.9 hours at 132.0 ng/mL | 91.4
  Participant 8: PET Scan 2, 5.0 hours at 304.0 ng/mL: number analyzed (Participants) | 1
  Participant 8: PET Scan 2, 5.0 hours at 304.0 ng/mL | 97.5
  Participant 8: PET Scan 3, 220.5 hours at 21.7ng/mL: number analyzed (Participants) | 1
  Participant 8: PET Scan 3, 220.5 hours at 21.7ng/mL | 53.9

34. Secondary Outcome: Trough of [18F]-IMA601
Time Frame: Day 1 up to Day 10
Population: Data for trough volume of distribution of [18F]-IMA601 was not collected and analyzed because steady state was not achieved due to non-periodic administration before the imaging sessions.
Arm/Group | Group 1: ASN51 Low Dose | Group 2: ASN51 High Dose
Number analyzed (Participants) | 0 | 0

35. Secondary Outcome: Receptor Occupancy as Assessed by Plasma Concentration That Corresponds to 50% Occupancy (EC50)
Description: Change in VT from baseline to post-dose scans were interpreted as an effect of O-GlcNAcase occupancy by ASN51. Occupancy estimates were plotted against plasma concentrations of ASN51, corresponding to the start of each post-dose PET scan. The following model was fitted to the occupancy data set: Occ=100*Cp/Cp+EC50. Where Occ was the target occupancy (%), Cp was measured plasma concentration of ASN51 (ng/ml) and EC50 was the plasma concentration of ASN51 that corresponds to 50% occupancy. Summarized data was reported for all participants.
Time Frame: Up to 220.5 hours post-dose on Day 1
Population: PET population included all participants in the safety population who had a baseline PET scan, at least 1 post-baseline PET scan, and a PK result immediately preceding a PET scan.
Measure: Mean (95% Confidence Interval); unit: ng/mL
Groups:
- ASN51: Participants received low and high doses of ASN51, orally, QD for 14 days in fasted or fed state.
Arm/Group | ASN51
Number analyzed (Participants) | 8
ng/mL | 17.6 [9.2 to 25.9]

ADVERSE EVENTS:
Time Frame: Baseline up to end of the study (approximately 4.5 months)
Description: Safety population included all participants who received at least one dose of the study drug.
Arm/Group | Group 1: ASN51 Low Dose | Group 2: ASN51 High Dose
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 4/6 | 3/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: ASN51 Low Dose (N=6) | Group 2: ASN51 High Dose (N=6)
Catheter site pain (General disorders) | 1 | 1
Catheter site related reaction (General disorders) | 1 | 1
Headache (Nervous system disorders) | 0 | 2
Lethargy (Nervous system disorders) | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Hordeolum (Infections and infestations) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-01-23): https://cdn.clinicaltrials.gov/large-docs/05/NCT05725005/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-13): https://cdn.clinicaltrials.gov/large-docs/05/NCT05725005/SAP_001.pdf